CLINICAL TRIAL: NCT00216788
Title: The Effect of Proton Pump Inhibitors on Transmucosal Esophageal Leak
Brief Title: The Effect of Nexium on Transmucosal Esophageal Leak
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Main Line Health (Other)
Collaborators: AstraZeneca (Industry); Sharpe-Strumia Research Foundation (Other); Cancer Research Foundation of America (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRUSESOM0388
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2005-11

CONDITIONS: Reflux; Esophagitis; Barrett's Esophagus
Keywords: Sucrose; Barrett's esophagus; Esophagitis; GERD; Reflux; Esophagus; Esomeprazole
MeSH Terms: conditions — Gastroesophageal Reflux; Esophagitis; Barrett Esophagus | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole (Nexium) 40 mg/day

SUMMARY:
In a related study, the investigators have found evidence that patients with Barrett's esophagus have a leak for oral sucrose to leave their upper gastrointestinal tract, enter the blood, and be filtered into urine. The amount of sucrose appearing in an overnight urine sample can be used to indicate the presence of Barrett's esophagus and/or esophagitis in a patient reporting with reflux (GERD) symptoms. The leak is presumably in the Barrett's epithelium itself. This phenomenon will be used to test if a standard 8 week therapy of Nexium in a first-time-presenting GERD patient can reduce the leak as a means of assessing the efficacy of the drug in that patient. The investigators predict that Nexium will reduce leak in esophagitis but not Barrett's patients.

DETAILED DESCRIPTION:
In a related study, we have found evidence that patients with Barrett's esophagus have a leak for oral sucrose to leave the lumen of their upper gastrointestinal tract, enter the blood, and be filtered into urine. Normally the disaccharide sucrose cannot leave the lumen of the gastrointestinal tract without being first hydrolyzed to glucose and fructose. Appearance of the disaccharide in the bloodstream suggests a paracellular leak of some type in the upper gastrointestinal tract. Once in the blood, sucrose is likewise not taken up or metabolized by the kidney but simply filtered into the urine. The amount of sucrose appearing in an overnight urine sample can be used to indicate the presence of Barrett's esophagus and/or esophagitis in a patient reporting with reflux (GERD) symptoms. The leak is presumably in the Barrett's epithelium itself. This phenomenon will be used to test if a standard 8 week therapy of Nexium in a first-time-presenting GERD patient can reduce the leak as a means of assessing the efficacy of the drug in that patient. We predict that Nexium will reduce leak in esophagitis but not Barrett's patients.

In this study, patients over 18 years of age presenting with GERD symptoms to a primary care physician, will be recruited after providing informed consent. Patients will perform a sucrose leak test the evening after their recruitment by drinking a solution of 100 gms of sucrose in 200 cc of water at bedtime, then collecting an overnight urine sample (8 hrs). Within 5 days the patient will undergo an upper endoscopy exam. The patient will then begin Nexium therapy (40 mg/day of Esomeprazole) for 8 weeks, taking the dose each morning before breakfast. After 8 weeks the patient will undergo a second sucrose leak test as described above. Urine sucrose will be determined by HPLC.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting to a general practitioner / internist with symptoms of GERD defined as:

* Heartburn - uncomfortable, rising, burning sensation behind the breastbone
* Regurgitation of gastric acid or sour contents into the mouth
* Chest pain atypical for cardiac ischemia and more suggestive of GERD
* Symptoms for more than three weeks with no concurrent use of PPI's or H-2 blockers during that time period
* A score greater than or equal to 5 on the AstraZeneca RDQ

Exclusion Criteria:

* Any patients presenting with alarm symptoms (GI bleeding, dysphagia, weight loss, abdominal mass, lymphadenopathy, or recurrent vomiting)
* Diabetes (type I or II)
* Renal insufficiency defined as creatinine >1.6
* Under 18 years of age
* Prior surgery on esophagus, stomach or duodenum
* History of gastric/duodenal ulcers
* History of H. pylori
* Known history of Barrett's esophagus (recruited to parallel study)
* On Coumadin or Heparin therapy
* Chronic upper abdominal pain more consistent with dyspepsia or other diagnoses
* Noncompliant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2006-01; Study Completion 2006-01 (Estimated)

PRIMARY OUTCOMES:
Urine sucrose level falls below 90 mg after 8 weeks of therapy

SECONDARY OUTCOMES:
Reduction of patient symptoms consistent with GERD

CONTACTS AND LOCATIONS:
Overall Officials: James M Mullin, Ph.D., Principal Investigator — Main Line Health
Locations (1):
- Lankenau Hospital, Wynnewood, Pennsylvania, United States

REFERENCES:
- See also: Related Info — http://www.pubmed.gov